CLINICAL TRIAL: NCT04245956
Title: Impact of Mitral Valve Regurgitation on Coronary Haemodynamics and the Instantaneous Effect of Transcatheter Mitral Valve Repair: The MitraFLOW Study
Brief Title: Impact of Mitral Regurgitation on Coronary Haemodynamics and Instantaneous Effect of Transcatheter Mitral Valve Repair
Acronym: MitraFLOW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrolment
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, IGLESIAS Juan Fernando, Medical Doctor, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-0000
Record Dates: First submitted 2019-07-17; First posted 2020-01-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Mitral Valve Insufficiency; Coronary Stenosis; Mitral Regurgitation; Coronary Artery Disease
Keywords: Mitral Regurgitation; MitraClip; iFR; Coronary microcirculation; Coronary hemodynamics
MeSH Terms: conditions — Mitral Valve Insufficiency; Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: MitraFLOW is a prospective, investigator-initiated, monocentric, open-label, non-randomized pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter Mitral Valve Repair arm (Experimental): Patients with severe Mitral Insufficiency with concomitant intermediate coronary artery stenosis undergoing Transcatheter Mitral Valve Repair using the percutaneous edge-to-edge MitraClip system
  Interventions: Procedure: Measure of hemodynamic indices in a stenosed coronary artery using a pressure wire

INTERVENTIONS:
Procedure: Measure of hemodynamic indices in a stenosed coronary artery using a pressure wire — The intervention consists of measuring a series of hemodynamic indices in a stenosed coronary using a pressure wire, immediately before and after transcatheter mitral valve repair using the percutaneous edge-to-edge MitraClip system in patients with severe mitral insufficiency and concomitant intermediate coronary artery stenosis.
  Other Names: MitraClip

SUMMARY:
In the present study, the investigators aim to use the in-vivo Transcatheter Mitral Valve Repair (TMVR) model to determine how Mitral Regurgitation (MR) affects coronary hemodynamics in patients affected with severe MR and concomittant angiographically-documented coronary artery disease. The investigators will also provide unique physiologic data on the acute effect of TMVR using the MitraClip system on coronary microcirculation in patients with severe MR.

DETAILED DESCRIPTION:
Consecutive patients with significant degenerative or functional MR planned for TMVR using the percutaneous edge-to-edge MitraClip system will be assessed for study eligibility. Patients with documented concomitant coronary artery disease, defined as coronary artery stenosis of 50% diameter or more in at least 1 epicardial coronary artery, will be informed about the study. Written informed consent will be obtained from all patients before enrolment in the study.

The TMVR procedure will be performed under general anesthesia with fluoroscopy and transesophageal echocardiographic guidance using the MitraClip device via a femoral venous approach. Cardiac catheterisation and coronary angiography will be undertaken via the transradial route, using standard equipment. The hemodynamic data listed below will be acquired immediately before and after TMVR.

For all lesions, intracoronary blood flow and pressure measurements will be used to generate the following intracoronary physiological parameters:

* Fractional Flow Reserve, FFR.
* Absolute coronary Blood Flow, ABF.
* Coronary Flow Reserve, CFR.
* Index for Microvascular Resistance, IMR.
* Baseline Resistance Index, BRI.
* Resistance Reserve Ratio, RRR.
* Instantaneous wave-free ratio, iFR

Post-procedural evaluation: Patients will be followed up according to local standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients with significant degenerative or functional MR planned for TMVR with the percutaneous edge-to-edge mitral valve repair MitraClip system;
3. Patients with ≥ 1 coronary artery lesion with angiographically-documented ≥50% diameter stenosis,
4. Patient willing and able to provide written informed consent.

Exclusion Criteria:

1. Previous coronary artery bypass surgery;
2. Presence of ≥1 coronary total occlusion(s);
3. Documented non-viable myocardium in the area of the corresponding coronary artery being studied;
4. Severe left ventricular systolic dysfunction (<30%);
5. Cardiogenic shock/hemodynamic instability at the time of intervention (heart rate<50 beats per minute, systolic blood pressure <90mmHg) and/or need for mechanical/pharmacologic hemodynamic support;
6. Systolic pulmonary artery pressure > 70 mmHg on baseline echocardiography;
7. Significant contraindication to adenosine administration (e.g. heart block, severe asthma);
8. Extremely calcified or tortuous vessels precluding invasive coronary physiology measurement;
9. Acute coronary syndrome with recent ST-elevation myocardial infarction <5 days prior to randomization, or ongoing non-ST elevation acute coronary syndrome with biomarkers (cardiac troponin) still rising;
10. Hypertrophic cardiomyopathy, restrictive pericarditis, constrictive pericarditis, infiltrative cardiomyopathy;
11. Participation or planned participation in another clinical trial, except for observational registries;
12. Patients unable or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Fractional Flow Reserve (FFR), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the Fractional Flow Reserve (FFR).
Change from baseline of instantanepous wave free ration (iFR), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the instantanepous wave free ration (iFR).
Change from baseline of Resting Full-Cycle Ratio (RFR), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the Resting Full-Cycle Ratio (RFR).
Change from baseline of Absolute coronary Blood Flow (ABF), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the Absolute coronary Blood Flow (ABF).
Change from baseline of Coronary Flow Reserve (CFR), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the Coronary Flow Reserve (CFR).
Change from baseline of the Index for Microvascular Resistance (IMR), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the Index for Microvascular Resistance (IMR).
Change from baseline of the Baseline Resistance Index (BRI), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the Baseline Resistance Index (BRI).
Change from baseline of the Resistance Reserve Ratio (RRR), after Transcatheter Mitral Valve Repair (TMVR). | Immediately post TMVR
  The primary endpoint of the study is the invasive pressure-derived physiological assessment of angiographically-documented intermediate coronary artery lesions before and after TMVR of the Resistance Reserve Ratio (RRR).

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland